CLINICAL TRIAL: NCT03508349
Title: Effectiveness of Intermittent Screening and Treatment of Malaria in Pregnancy (ISTp) on Maternal and Birth Outcomes in Selected Districts in Rwanda
Brief Title: Routine Antenatal Care Versus Screening and Treatment of Malaria in Pregnancy in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Rwanda Malaria and Other Parasitic Diseases Division (MOPDD) (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6829
Record Dates: First submitted 2018-01-23; First posted 2018-04-25 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Malaria in Pregnancy

STUDY DESIGN:
Intervention Model Description: Health facilities in high malaria transmission zones were pair matched and then randomized to be an intervention or a control facility.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IST using RDT (Experimental): Women presenting for their first ANC visit to facilities will be consecutively enrolled after providing informed consent. Women in the intervention group (IST+ routine care) will be tested for malaria at the health center during their ANC visits with an RDT. If positive, they will be treated with artemisinin-based combination therapy (ACT) in second or third trimester or quinine in the first trimester.
  Interventions: Diagnostic Test: IST
- Routine Antenatal Care (No Intervention): Women presenting for their first ANC visit to facilities will be consecutively enrolled after providing informed consent. Women in the comparison group (routine care) will receive routine antenatal care services per the national guidelines. They will not be tested for malaria at each antenatal care visit unless they are symptomatic for malaria.

INTERVENTIONS:
Diagnostic Test: IST — Women in the control group will receive routine care, which does not include testing for malaria with a rapid diagnostic test unless symptomatic for malaria. Women in the intervention group will receive this additional testing for malaria at each antenatal care, regardless of whether she is symptomatic for malaria.
  Arms: IST using RDT

SUMMARY:
The main aim of this study is to test the primary hypothesis that the addition of intermittent screening and treatment of malaria in pregnant women (ISTp) who receive routine antenatal care (ANC) in health facilities in high malaria transmission areas in Rwanda will reduce malaria prevalence among pregnant women when compared to routine antenatal cares services alone.

DETAILED DESCRIPTION:
More specifically, the primary objective is to understand the effect of ISTp in a context where routine antenatal care does not include malaria chemoprohylaxis and whether this intervention is protective against malaria during pregnancy. The secondary objective is to determine whether this intervention results in an improvement in other key maternal and newborn health outcomes including maternal anemia, low birth weight and prematurity. The third objective is to determine the feasibility, effectiveness and acceptability of ISTp among women who receive ISTp and among health workers who deliver this intervention.

This study will establish if testing and treating pregnant women is effective, feasible and whether it adds an additional burden to the work already being undertaken by facility-based health workers who provide antenatal care services. It is expected that the study will result in information to develop appropriate approaches that can be implemented in Rwanda in the prevention of malaria in pregnancy in addition to the use of preventive measures such as insecticide treated mosquito nets (ITNs) and case management. This information may potentially also be used by other countries with similar patterns of malaria transmission.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 or older who have their first ANC visit during the study recruitment period
* Willing to participate

Exclusion Criteria:

* • Pregnant women below the age of 18

  * Not willing to participate

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant at the time of enrollment in the study
Enrollment: 1786 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of placental malaria at delivery (tested by PCR) | at the time of delivery
  comparison of prevalence of malaria between women in intervention and control sites

SECONDARY OUTCOMES:
Prevalence of maternal anemia at delivery | at the time of delivery
  comparison of prevalence of maternal anemia between women in intervention and control sites
Prevalence of low birth weight babies (<37 weeks gestation) | at the time of delivery
  comparison of prevalence of LBW between women in intervention and control sites
Prevalence of preterm births | at the time of delivery
  comparison of prevalence of preterm births between women in intervention and control sites
Episodes of clinical malaria during the course of the pregnancy | assessed at the time of delivery
  description of the number of episodes of malaria detected during antenatal care visits during pregnancy

OTHER OUTCOMES:
Adverse outcome of pregnancy - abortions, still births and neonatal deaths | assessed at the time of delivery
  Description of the number of adverse outcomes by group

CONTACTS AND LOCATIONS:
Overall Officials: Reena Sethi, DrPH, Principal Investigator — Jhpiego
Locations (14):
- Rwanda (14):
  - Busoro-Gishamvu Health Center, Huye, South
  - Huye Police Health Center, Huye, South
  - Maraba Health Cente, Huye, South
  - Mukura Health Center, Huye, South
  - Rango Health Center, Huye, South
  - Rubona Health Center, Huye, South
  - Rwaniro, Huye, South
  - Sovu Health Center, Huye, South
  - Kamonyi Health Center, Kamonyi, South
  - Kayenzi Health Center, Kamonyi, South
  - Mugina Health Center, Kamonyi, South
  - Musambira Health Center, Kamonyi, South
  - Nyagihamba Health Center, Kamonyi, South
  - Nyamiyaga Health Center, Kamonyi, South

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alruwaili M, Uwimana A, Sethi R, Murindahabi M, Piercefield E, Umulisa N, Abram A, Eckert E, Munguti K, Mbituyumuremyi A, Gutman JR, Sullivan DJ. Peripheral and Placental Prevalence of Sulfadoxine-Pyrimethamine Resistance Markers in Plasmodium falciparum among Pregnant Women in Southern Province, Rwanda. Am J Trop Med Hyg. 2023 Oct 2;109(5):1057-1062. doi: 10.4269/ajtmh.23-0225. Print 2023 Nov 1. PMID 37783456
- [Derived] Uwimana A, Sethi R, Murindahabi M, Ntirandeka C, Piercefield E, Umulisa N, Abram A, Eckert E, Munguti K, Sullivan D, Uyizeye D, Mbituyumuremyi A, Gutman JR. Effectiveness of Intermittent Screening and Treatment of Malaria in Pregnancy on Maternal and Birth Outcomes in Selected Districts in Rwanda: A Cluster Randomized Controlled Trial. Clin Infect Dis. 2023 Jul 5;77(1):127-134. doi: 10.1093/cid/ciad128. PMID 36896967